CLINICAL TRIAL: NCT01816737
Title: Fetal Blood Flow Response to Partial Occlusion by External Compression
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC13191-12CTIL; 0191-12-MMC (Other: Helsinki committee , MeirMc, Israel)
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Gestational Age

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Two earlier studies showed measurable fetal hemodynamics changes caused by external pressure induced by te abdominal ultrasound transducer. The investigators would like to study the response of flow in main fetal vessels to different, mild to moderate pressures induced by the abdominal transducer. The pressure induced by the transducer will be measured by a digital computed manometer. The flow chances in fetal vessels will be measured by ultrasound Doppler. Measurements will be taken on different pregnancy weeks, on one occasion in each pregnant woman. Ones without applying transducer pressure (control) and ones after applying mild pressure.

ELIGIBILITY:
Inclusion Criteria:

singleton

Exclusion Criteria:

multiple gestation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
pulsatility index in fetal vessels | at the time of pressure aplication